CLINICAL TRIAL: NCT06519448
Title: Reducing Non-Alcoholic Steatohepatitis Study
Brief Title: Reducing Non-Alcoholic Steatohepatitis
Acronym: RedNASH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Petr Hribek, Principal Investigator, Military University Hospital, Prague
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RedNASH
Record Dates: First submitted 2024-07-03; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Non-alcoholic Steatohepatitis; Liver Diseases; Diabetes Mellitus, Type 2; Fibrosis, Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Diabetes Mellitus, Type 2; Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NASH (Experimental): Patients with histological proven NASH (either diabetics and non-diabetics).
  Interventions: Drug: Empagliflozin 10 miligrams (mg)

INTERVENTIONS:
Drug: Empagliflozin 10 miligrams (mg) — Use of empagliflozin 10 mg daily for 12 months.

SUMMARY:
The goal of this clinical trial is to learn if empagliflozin works to treat non-alcoholic steatohepatitis in adults. The objectives are:

Primary Objective To evaluate the change in histological grading and staging of NASH in patients with confirmed non-alcoholic steatohepatitis (NASH) treated with empagliflozin for a duration of 48 weeks.

Secondary Objective To evaluate the change in findings from non-invasive liver elasticity measurements, laboratory tests, and anthropometric assessments after 48 weeks of empagliflozin administration.

Participants will:

Take empagliflozin every day for 12 months. Visit the clinic according to a protocol at weeks: 1, 2, 4, 12, 24, 36, 48 Visits includes checkups and tests (blood count, basic biochemistry, glycosylated hemoglobin, anthropometry, non-invasive liver stiffness measurement).

ELIGIBILITY:
Inclusion Criteria:

* Ability and eligibility to provide informed consent.
* Age between 18 and 75 years at the time of study initiation.
* Confirmed or excluded diagnosis of type 2 diabetes mellitus (DM2) according to the target group (OGTT test, HbA1c).
* Diagnosis of NASH confirmed by a central pathologist based on histological evaluation of a liver biopsy performed within 3 months prior to the initiation of the investigational drug. - The evaluation must include determination of the process activity according to the NAFLD Activity Score (NAS).
* HbA1c value ≤ 80 mmol/mol.
* For women of childbearing potential, willingness to use at least two adequate methods of contraception.

Exclusion Criteria:

* Contraindication to liver biopsy.
* Documented episode of ketoacidosis.
* Contraindication or hypersensitivity to empagliflozin.
* Presence of acute or chronic illness that, in the investigator's opinion, could jeopardize the health or safety of the patient.
* HbA1c value > 80 mmol/mol.
* Inability to safely discontinue thiazolidinedione (pioglitazone) therapy.
* Liver disease of other etiologies, including viral hepatitis B and C, autoimmune hepatitis, alpha-1 antitrypsin deficiency, hemochromatosis, Wilson's disease, primary sclerosing cholangitis, primary biliary cholangitis, or liver cirrhosis (Child-Pugh A, B, C) of any etiology.
* Use of medications or medical procedures that induce liver steatosis or fibrosis.
* Proven alcohol use exceeding: Men > 30 g/day, Women > 20 g/day.
* History of acute or chronic pancreatitis.
* Known dependence on or use of illegal addictive substances.
* Significant weight gain or loss: +/- 10% in the last three months.
* Diagnosis of malignant disease (except treated benign or skin tumors) in the last 5 years.
* Stroke or myocardial infarction in the last 6 months.
* Clinically significant dyspnea New York hear association (NYHA) grade III or higher.
* Proven heart failure with a left ventricular ejection fraction below 40%.
* estimated glomerular filtration rate(eGFR) values lower than 30 ml/min/1.73 m² or creatinine clearance lower than 30 ml/min.
* Proven diabetic foot syndrome requiring amputation or with an existing defect.
* Planned pregnancy, ongoing lactation or pregnancy, positive pregnancy test, lack of at least two adequate contraceptive methods in women of childbearing potential.
* Participation in another interventional study within the last 3 months before study entry.
* Legal incapacity or reduced ability to perform legal acts.
* Serving a prison sentence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in histological activity after 12-month treatment with empagliflozin | 12 months
  Non-alcoholic Fatty Liver Disease Activity Score (NAS) change after intervention. The NAS can range from 0 to 8 and is calculated by the sum of scores of steatosis (0-3), lobular inflammation (0-3) and hepatocyte ballooning (0-2). In patients with NAFLD, NAS score of ≥ 5 strongly correlated with a diagnosis of "definite NASH" whereas NAS ≤ 3 correlated with a diagnosis of "not NASH".

SECONDARY OUTCOMES:
Change of liver stiffness | 12 months
  Liver stiffness measured in kilopascals (kPa) by transient elastography at baseline and after intervention.
Change of liver steatosis | 12 months
  Continuous attenuation parameter measured in decibels per meter (dB/m) at baseline and after intervention.
Anthropometry (body weight) | 12 months
  Measurement of body weight measured in kilograms (kg) and change from baseline.
Anthropometry (height) | 12 months
  Measurement of body height measured in metres (m) to calculate Body Mass Index (BMI).
Anthropometry (BMI) | 12 months
  Change in BMI from baseline (measured in kg/m^2).
Liver functional tests | 12 months
  Change in activity liver functional tests (LFT) all measured in microkatals per liter (ucat/L) from baseline.
  These tests comprise:
  Alanine transaminase (ALT) Aspartate transaminase (AST) Gamma-glutamyl transferase (GGT) Alkaline phosphatase (ALP)
Bilirubin level | 12 months
  Change in activity concentration of bilirubin measured in micromoles per liter (umol/L) from baseline.
Lipidogram | 12 months
  Change in cholesterol, LDL cholesterol, HDL cholesterol, triglycerides (measured in mmol/L) from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Military Hospital, Prague, Czechia